CLINICAL TRIAL: NCT04800939
Title: The Effect of Acupressure on the Sleep Quality and Daytime Sleepiness of Surgical Nurses During the COVID-19 Pandemic Process
Brief Title: The Effect of Acupressure on the Sleep Quality and Daytime Sleepiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Mersin Uni
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sleep
Keywords: Acupressure; placebo acupressure; nurses; sleep quality; daytime sleepiness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: According to the randomization table, the information showing the nurses included in the research sample is assigned to the A and B groups will be put in an opaque envelope. This envelope will be kept by the coordinator researcher (GAU) when the researcher (TÇY), who has an acupressure application certificate, goes to the nurse's application. After filling out the "Informed Consent Form," he will open the envelope and learn which group the nurse is in. Since all nurses included in the study will be applied to the compression point, the participants will be blinded because they do not know that they are a study or control group. The researcher (TÇY), on the other hand, cannot be blinded due to the nature of the research. A statistician will analyze the data, and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure Group (Experimental): The experimental group will be given acupressure on their own, three times a week for four weeks, one hour before going to bed at night.
  Interventions: Other: Acupressure
- Placebo Acupressure Group (Other): The control group will be given plasebo acupressure on their own, three times a week for four weeks, one hour before going to bed at night.
  Interventions: Other: Plasebo acupressure

INTERVENTIONS:
Other: Acupressure — The experimental group will start with HT7 points and continue with SP6 points. The application will be carried out by determining the priority order of the points with the draw. Attention will be paid to the intensity and duration of the pressure deemed appropriate. Since the individuals' responses will differ, the stiffness and pressure will be adjusted according to the individual's sensitivity not to cause tissue damage. Before starting the application, around the area to be pressed for 20-30 seconds will be gently rubbed with palm. With the gentle rubbing of the surrounding tissue, the tension and tissue sensitivity in warming, relaxing and preparatory will be reduced, and the tissue will be relieved. After, the point determined will be pressed manually for 2 minutes.
  Other Names: Acupress
  Arms: Acupressure Group
Other: Plasebo acupressure — In the control group, the application will start with the points 1.5 cm around the HT7 and SP6 points. The application process will continue in the same way with acupressure group and the pressure intensity will be less.
  Other Names: Acupress
  Arms: Placebo Acupressure Group

SUMMARY:
This randomized controlled trial evaluates the effect of acupressure application on nurses' sleep quality and daytime sleepiness providing care in surgical clinics. This study hypothesizes that acupressure improves sleep quality and reduces daytime sleepiness.

DETAILED DESCRIPTION:
Methods: In the study, 60 nurses were randomly assigned to acupressure and placebo acupressure groups. To the acupressure group (n = 30), an average of 10 minutes will be applied to the Shen Men, the 7th acupoint (HT7) of the heart meridian located between the ulna and pisiform bones, on the radial side of the flexor carpi ulnaris tendon, and the Sanyinjia points on the splenic meridian (SP6) located on the inner side of the lower leg, four fingers above the ankle and behind the tibia. In the placebo acupressure group (n = 30), the points 1.5 cm away from the HT7 and SP6 points (four points in total) will be applied for an average of 10 minutes. The primary outcome of the research is the effect of acupressure on the sleep quality of nurses. The secondary outcome of the study is to determine the effect of acupressure on daytime sleepiness. The outcomes will be collected before and four weeks after the acupressure and placebo acupressure administration.

ELIGIBILITY:
Inclusion Criteria:

The experimental group criteria to be included in the study;

* Caring for COVID-19 patients during the research,
* Working in surgery services before the pandemic,
* Agree to participate in the survey (those who signed the Informed Consent Form),
* Do not have physical problems that prevent acupressure application to HT7 (wrist) and SP6 (over four fingers of the ankle) points,
* No experience of acupressure,
* Not diagnosed with sleep disorder and not receiving medical treatment,
* No coffee, cigarette, and alcohol addiction,
* No mental illness,
* Working in the night shift,
* Don't work more than three-night shifts a week.

The control group criteria to be included in the study;

* Caring for COVID-19 patients during the research,
* Working in surgery services before the pandemic,
* Agree to participate in the survey (those who signed the Informed Consent Form),
* Do not have physical problems that prevent acupressure application to points 1.5 cm away from HT7 (wrist) and SP6 (4 fingers above the ankle) points,
* No experience of acupressure,
* Not diagnosed with sleep disorder and not receiving medical treatment,
* No coffee, cigarette, and alcohol addiction,
* No mental illness,
* Working in the night shift,
* Do not work more than three-night shifts a week.

Exclusion Criteria:

The experimental group criteria not to be included in the study;

* Do not care for COVID-19 patients during the research,
* Do not work in surgery services before the pandemic,
* Do not agree to participate in the study,
* Having physical problems that prevent acupressure application to HT7 (wrist) and SP6 (over four fingers of the ankle) points,
* Diagnosed with sleep disorder and receiving medical treatment,
* Using drugs that cause sleep problems (antidepressants, analgesics, beta-adrenoreceptor antagonists, dopamine agonists, etc.),
* Addicted to coffee, cigarette, and alcohol,
* With mental illness,
* Working more than three-night shifts a week,
* Working on a fixed day shift.

The control group criteria not to be included in the study;

* Do not care for COVID-19 patients during the research,
* Do not work in surgery services before the pandemic,
* Do not agree to participate in the study,
* Having physical problems that prevent acupressure application to points 1.5 cm away from HT7 (wrist) and SP6 (4 fingers above the ankle) points,
* Diagnosed with sleep disorder and receiving medical treatment,
* Using drugs that cause sleep problems (antidepressants, analgesics, beta adrenoreceptor antagonists, dopamine agonists, etc.),
* Addicted to coffee, cigarette, and alcohol,
* With mental illness,
* Working more than three-night shifts a week,
* Working on a fixed day shift.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Sleep quality evaluated using the Pittsburgh Quality Sleep Index | Change from before implementation and 4th week of practice.
  The total scale score is in the range of 0 (minimum) -21 (maximum), and the high total Pittsburgh Quality Sleep Index (PSQI) score indicates that sleep quality is low. A total PSQI score between 0-4 indicates good sleep quality, while between 5-21 shows that sleep quality is low.

SECONDARY OUTCOMES:
Daytime sleepiness evaluated using the Epworth Sleepiness Scale | Change from before implementation and 4th week of practice
  This scale, which is a four-point Likert type, aims to evaluate the probability of sleepiness during the individual's daily life between 0-3 points. The scale score is in the range of 0 (minimum) -24 (maximum), and a total Epworth Sleepiness Scale score of 11 or above indicates excessive daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Altun Ugras, Doctorate, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No